CLINICAL TRIAL: NCT00337116
Title: Intravenous Isosorbide Dinitrate Versus Sublingual Isosorbide Dinitrate for the Relief of Acute Anginal Episodes in Acute Coronary Syndrome (ACS) Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: LOGISTIC DIFFICULTIES
Sponsor: Soroka University Medical Center (Other)
Responsible Party: DORON ZAHGER, SOROKA UNIVERSITY MEDICAL CENTER
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: sor435006ctil
Record Dates: First submitted 2006-06-14; First posted 2006-06-15 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2007-01

CONDITIONS: Unstable Angina; Myocardial Infarction
MeSH Terms: conditions — Angina, Unstable; Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: iso sorbide dinitrate iv bolus or s/l

SUMMARY:
This is a randomized, double blind, placebo-controlled study, clinical trail designed to evaluate the efficacy safety and superiority of intravenous boluses of isosorbide dinitrate for the relief of acute anginal pain episodes in acute coronary syndrome patients in comparison with the usual manner of S/L isosorbide dinitrate .

DETAILED DESCRIPTION:
Analgesia is an important element in the management of ACS patients. Pain contributes to the heightened sympathetic activity that is particularly prominent during periods of acute STEMI, NSTEMI and unstable angina and consequentially causes elevation of tissue oxygen demand. Control of cardiac pain is typically accomplished with a combination of oxygen, analgesic (e.g. morphine) beta blockers agents and primarily nitrates.

Sublingual nitrates are currently the guidelines recommended preparation for instant relief of brief episodes of pain. In patients with prolonged periods of waxing and waning chest pain, drip of intravenous nitrates may be of benefit in controlling of symptoms and correcting ischemia.

Intravenous nitrates are also indicated for the treatment of acute decompensated CHF patients with pulmonary edema, nevertheless the current treatment for these patients edema is repeated intravenous boluses of and not sublingual isosorbide dinitrate, followed by continuous drip. Although there is no hard data on intravenous high-dose nitrates for the relief of acute anginal pain episodes, our clinical impression with this method is excellent.

Intravenous boluses of isosorbide dinitrate in a hospital setting provides immediate, accurate (bioavailability ) and is an easily controlled modality for providing nitrates.

Since intravenous boluses of isosorbide dinitrate is the standard care for acute anginal pain episodes in our ICCU at this time, a well designed comparative study for the two methods would help it to become a guideline and not a matter of choice in these cases.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years or older.
2. Admission to the ICCU with ACS (non-ST elevation acute coronary syndrome or 24 hours after ST elevation myocardial infarction) .
3. Presence of ischemic symptoms (≥5 minutes) during hospitalization.
4. Pain assessment of 3 out of 10 on Visual Analog Scale (VAS) 1 or dynamic ECG findings (ST segment deviation ≥0.05 mV or T wave inversion ≥ 0.3 mV)
5. Willing and able to provide written informed consent according to the regulations of the Ministry of Health and the Helsinki committee instructions.

   -

Exclusion Criteria:

1. Patient who meet any of the following criteria are excluded from the study:
2. Persistent ST-segment elevation ≥ 1 mV in 2 or more contiguous leads or new LBBB.
3. Acute pulmonary edema
4. Sepsis
5. Sustained systolic blood pressure < 90 mm Hg or evidence of cardiogenic shock
6. Pregnant women
7. Use at randomization of agents known to enhance the efficacy of nitrates.
8. Clinically significant aortic stenosis
9. Cr > 2 mg/dL
10. Participation in another trial of an investigational drug or device on randomization.
11. Allergy or sensitivity to nitatrate compounds
12. Acute episode of cerebrovascular attack
13. Inability to comply with the protocol and follow-up

    -

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: doron zahger, prof, Principal Investigator — soroka university medical center israel
Locations (1):
- Intensive Cardiac Care Unit, Beersheba, Israel